CLINICAL TRIAL: NCT00829231
Title: Open Label, Phase 1 to Evaluate the Effect of Hepatic Impairment on the Pharmacokinetic of Sorafenib ( BAY43-9006)
Brief Title: Hepatic Impairment Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12349
Record Dates: First submitted 2009-01-23; First posted 2009-01-26 (Estimated); Last update posted 2014-11-03 (Estimated); Status verified 2014-10

CONDITIONS: Liver Disease
Keywords: Liver disease
MeSH Terms: conditions — Liver Diseases | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Experimental)
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006)
- Arm 2 (Experimental)
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006)
- Arm 3 (Experimental)
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006)

INTERVENTIONS:
Drug: Sorafenib (Nexavar, BAY43-9006) — Mildly Hepatic Impaired Subjects
  Arms: Arm 1
Drug: Sorafenib (Nexavar, BAY43-9006) — Moderately Hepatic Impaired Subjects
  Arms: Arm 2
Drug: Sorafenib (Nexavar, BAY43-9006) — Healthy Subjects
  Arms: Arm 3

SUMMARY:
This study is to find out how the subject's body processes and reacts to the study drug, and to find out how long it remains in the subjects system after one dose. Subjects with varying degrees of liver function are being asked to participate in this study. Study results from subjects with normal liver function will be compared with study results from subjects with impaired liver function.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Subjects, Child Pugh A and Child Pugh B Liver Disease Patients.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2009-01; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
PK measurements | Day 1-6

SECONDARY OUTCOMES:
Physical Exam | Screening, Day 6
Labotatory Safety, Chemistry panel, PTT, hematology Urine Analysis | Screening Day 1, Day 6
ECG | Screening Day 1, Day 6
Vital Signs | Screening Day 1, Day 6
Follow up phone call | Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (3):
- United States (3):
  - Miami, Florida
  - Orlando, Florida
  - Knoxville, Tennessee